CLINICAL TRIAL: NCT03632629
Title: Treatment Effects of Cognitive Training on Children With Attention Deficit Hyperactivity Disorder and Developmental Delay
Brief Title: Effects of Cognitive Training on Children With Attention Deficit Hyperactivity Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Ru-Lan Hsieh, Principal investigator, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018SKHADR028
Record Dates: First submitted 2018-07-13; First posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: cognitive training; developmental delay; children; therapeutic effect
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Learning Disabilities

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Active Comparator): 3 months of individualized interactive cognitive training, 2 times per week, 15 min per session, a total of 24 sessions, in addition to traditional rehabilitation programs.
  Interventions: Other: interactive cognitive training
- control group (No Intervention): 3 months of traditional rehabilitation programs, without individualized interactive cognitive training.

INTERVENTIONS:
Other: interactive cognitive training — Using interactive brain club system training to children with attention deficit hyperactivity disorder with developmental delay
  Arms: study group

SUMMARY:
Using a single blind, randomized controlled design to study the additional therapeutic effects of cognitive training on traditional rehabilitation programs for children with attention deficit hyperactivity disorder and developmental delays.

DETAILED DESCRIPTION:
A total of 30 children with attention deficit hyperactivity disorder and developmental delays who are receiving traditional rehabilitation programs will be enrolled.

The participants will be randomized into two groups, including study group (traditional rehabilitation program with additional cognitive training: 2 times per week, 15 min per session, a total of 24 sessions) and control group (traditional rehabilitation program without additional cognitive training).

Memory related functions, quality of life, and physical function evaluations will be performed at baseline, 3 months and 6 months later, respectively.

Evaluator will be blinded to the group's classification during the whole course of study.

ELIGIBILITY:
Inclusion Criteria:

* children diagnosed with attention deficit hyperactivity disorder with developmental delay receiving regular rehabilitation programs intelligence quotient 70 or greater

Exclusion Criteria:

* age less than 4 years or elder than 8 years children diagnosed with attention deficit hyperactivity disorder receiving regular rehabilitation programs intelligence quotient less than 70

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
change of attention | scores change from baseline to 3 months of treatment, and 3 months after treatment
  score assessed by Swanson, Nolan and Pelham questionnaire

SECONDARY OUTCOMES:
change of visual motor integration | scores change from baseline to 3 months of treatment, and 3 months after treatment
  score assessed by Beery-Buktenica Visual Motor Integration Test
change of sensory integration | scores change from baseline to 3 months of treatment, and 3 months after treatment
  score assessed by Sensory Profile questionnaire
change of intelligence | scores change from baseline to 3 months of treatment, and 3 months after treatment
  score assessed by Wechsler Intelligence Scale for Children, including verbal, performance and total scores, the average score is 100, with higher scores indicating higher than average intelligence and lower scores indicating lower levels of intelligence
change of functional performance | changes from baseline to 3 months of treatment, and 3 months after treatment
  score assessed by Pediatric Outcome Data Collection Instrument
change of health-related quality of life | changes from baseline to 3 months of treatment, and 3 months after treatment
  score assessed by Pediatric Quality of Life Inventory-Generic Core Scales, including physical, psychosocial, and total scores, with higher scores representing better health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Lan Hsieh, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No